CLINICAL TRIAL: NCT04143659
Title: A Phase I Study to Evaluate the Pharmacokinetic and Pharmacodynamic Profile of Intramuscular or Subcutaneous Injections of Levonorgestrel Butanoate (LB) for Female Contraception
Brief Title: A Study to Evaluate the PK and PD of IM or SQ Injections of Levonorgestrel Butanoate (LB) for Female Contraception
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Clint Dart, Senior Program Director, NICHD, Premier Research
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CCN021
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Healthy Women; Female Contraception
MeSH Terms: interventions — levonorgestrel butanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LB injection 40mg intramuscular (IM) with 20 mg/ml concentration (Experimental): 27 subjects (18 with BMI <30mg^2; 9 with BMI >=30kg/m^2 and <40kg/m^2) were administered a single dose of levonorgestrel butanoate (LB) injection 40mg intramuscular (IM) using 20 mg/ml concentration
  Interventions: Biological: levonorgestrel butanoate (LB) injection
- LB injection 40 mg subcutaneous (SC) with 20 mg/ml concentration (Experimental): 32 subjects (25 with BMI <30mg^2; 7 with BMI >=30kg/m^2 and <40kg/m^2) were administered a single dose of levonorgestrel butanoate (LB) injection 40mg subcutaneous (SC) using 20 mg/ml concentration
  Interventions: Biological: levonorgestrel butanoate (LB) injection
- LB injection 50mg subcutaneous (SQ) with 70 mg/ml concentration (Experimental): 8 subjects (8 with BMI <40 kg/m2) will be administered a single dose of levonorgestrel butanoate (LB) injection 50mg intramuscular (IM) using 70 mg/ml concentration
- LB injection 60mg Subcutaneous (SQ) with 70 mg/ml concentration (Experimental): 32 subjects (16 with BMI <30mg^2; 16 with BMI >=30kg/m^2 and <40kg/m^2) will be administered a single dose of levonorgestrel butanoate (LB) injection 60mg subcutaneous (SC) using 70 mg/ml concentration
- LB injection 40 mg subcutaneous (SQ) with 70 mg/ml concentration (Experimental): 32 subjects (21 with BMI <30mg^2; 11 with BMI >=30kg/m^2 and <40kg/m^2) were administered a single dose of levonorgestrel butanoate (LB) injection 40mg subcutaneous (SC) using 70 mg/ml concentration
  Interventions: Biological: levonorgestrel butanoate (LB) injection

INTERVENTIONS:
Biological: levonorgestrel butanoate (LB) injection — The initial formulation of the investigational product (IP) is LB Injectable Suspension at a concentration of 40 mg/2 mL (20 mg/mL). Each vial contains 2 mL at 20mg/mL for a total of 40 mg. This formulation will only be used for dosing groups A and B with the injections completed as 40 mg IM (2 mL) or 40 mg SQ (2 mL).
  The second formulation of the investigational product (IP) is LB Injectable Suspension is a concentration of 140 mg/2 mL (70 mg/mL). Each vial contains 2 mL at 70 mg/mL for a total of 140 mg. This formulation will only be used for dosing groups B2, C, and D with the injections completed as 40 mg SQ (0.57 mL), 50 mg SQ (0.71 mL), and 60 mg SQ (0.86 mL).
  Arms: LB injection 40 mg subcutaneous (SC) with 20 mg/ml concentration; LB injection 40 mg subcutaneous (SQ) with 70 mg/ml concentration; LB injection 40mg intramuscular (IM) with 20 mg/ml concentration

SUMMARY:
This is a Phase I multicenter, open-label, dose-ranging, three-dose PK and PD study of injectable LB administered as an IM or SQ injection at 40 mg, and subsequently at 50mg SQ and then 60 mg SQ depending on the preliminary pharmacokinetic and pharmacodynamic results obtained with 40 mg dosing.

DETAILED DESCRIPTION:
This is a Phase I multicenter, open-label, dose-ranging, three-dose PK and PD study of injectable LB administered as an IM or SQ injection at 40 mg, and subsequently at 50 mg SQ and then 60 mg SQ depending on the preliminary pharmacokinetic and pharmacodynamic results obtained with 40 mg dosing.

Healthy normal weight and healthy obese women will be enrolled and followed as outpatients until return to ovulation and normal menses. The participation time is estimated to be approximately nine months. During this study, subjects will undergo a screening period prior to enrollment to confirm normal ovulatory function, and then receive active treatment with injection of LB administered via IM or SQ injection. A dose of LB administered IM (40 mg) or SQ (40 mg) was selected for initial evaluation for this study. Subjects will undergo frequent study and safety evaluations and will have serum samples taken to evaluate drug levels and ovulatory function, in addition to a transvaginal ultrasound (TVUS) at selected visits. Follow-up will continue until normal ovulatory cycles resume. Based upon detailed studies in non-human primates and our experience with the 40mg dose groups, it is expected that most subjects will resume menstrual cycles within 12 - 26 weeks after the injection. Subjects will continue to be followed for one normal cycle after the return of menses.

This dose-ranging, PK/PD study will be conducted at seven of the female Contraceptive Clinical Trials Network (CCTN) sites in the U.S. and will enroll approximately 136 women who demonstrate normal ovulatory function during the baseline cycle. Enrollment will be stratified to target that 50% of the subjects have a BMI >30 kg/m^2 and <40 kg/m^2 and approximately 50% of subjects have a BMI <30 kg/m^2 in each dose group.

LB injections will be administered at the study site by a trained research nurse or physician. The SQ injections should be done slowly under the skin in the abdomen to ensure drug is dispensed into the tissue layer between the skin and the muscle following standard procedures for subcutaneous injections. For IM injections, the staff should inject LB slowly in the deltoid avoiding the injection into blood vessels following standard procedures for intramuscular injections. (The SQ injection may be given in a different location than the abdomen and the IM injection in a different location than the deltoid with the approval of the Medical Monitor.) The study subject will be observed for at least 30 minutes after the injection before release from the study site.

The different combinations of doses and methods of administration (IM or SQ) will be given in sequential stages, using two different LB concentrations (20 mg/mL or 70 mg/mL) as described below.

Enrollment Stage A: 40 mg IM with 20 mg/ml concentration (27 subjects [18 with BMI <30 kg/m^2; 9 with BMI >30 kg/m^2 and <40 kg/m^2])

Enrollment Stage B: 40 mg SQ with 20 mg/ml concentration (32 subjects [25 with BMI <30 kg/m^2; 7 with BMI >30 kg/m^2 and <40 kg/m^2])

Enrollment Stage B2: 40 mg SQ with 70 mg/ml concentration (32 subjects [21 with BMI <30 kg/m^2; 11 with BMI >30 kg/m^2 and <40 kg/m^2])

Enrollment Stage C: 50 mg IM with 70 mg/ml concentration (8 subjects [8 with BMI <40 kg/m^2])

Enrollment Stage D: 60 mg SQ with 70 mg/ml concentration (32 subjects [16 with BMI <30 kg/m^2; 16 with BMI >30 kg/m^2 and <40 kg/m^2])

Stages will be performed sequentially; PK/PD assessments will be performed. The target numbers for enrollment in each BMI category are approximate.

Results of the preliminary pharmacokinetic and pharmacodynamic results for the three 40 mg dose groups support moving forward with a maximum dose of 60 mg rather than 70 mg SQ. However, after reviewing these results, the FDA recommended a SAD study with a 50 mg SQ dose before proceeding with 60 mg LB administered SQ. The following enrollment table reflects groups for this revised protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health with no chronic medical conditions that result in periodic exacerbations that require significant medical care.
2. Age between 18 and 40 years inclusive at the injection visit.
3. BMI < 40 kg/m2.
4. Intact uterus with at least one ovary.
5. Pap test within ASCCP or ACOG guidelines such that additional treatment will not be required during the study period. If a copy of a Pap test (and indicated follow-up testing) is not available and the subject is 21 years or older, a Pap test should be done during the screening period.
6. Regular menstrual cycles that occur every 21-35 days:

6a. If subject is postpartum or post-second trimester abortion, she must have 3 menses (2 cycles) prior to enrollment.

6b. If subject had a first trimester abortion or pregnancy loss, she must have one spontaneous menses prior to enrollment.

7. Have a negative urine pregnancy test at the injection visit and no unprotected heterosexual intercourse for the previous 10 days.

8. Not at risk for pregnancy for the duration of study participation (screening through last phone contact), defined as one of the following: 8a. heterosexually abstinent; 8b. previous female permanent contraception procedure; 8c. in a monogamous relationship with a vasectomized partner; 8d. consistent use of a non-hormonal barrier method with every act of intercourse (e.g. condoms or diaphragm + spermicide).

8e. use copper IUD 9. Subjects must be ovulatory as confirmed by a documented screening progesterone (P4) level ≥ 3 ng/ml by local laboratory.

10. In the opinion of the investigator, subject is willing and able to comply with the protocol requirements.

11. Willing to record requested information in the daily diary. 12. Lives within the study site catchment area or within a reasonable distance from the site.

13. Understands and signs an Institutional Review Board (IRB) approved informed consent form prior to undergoing any screening assessments (including fasting blood draw).

14. Agrees not to participate in any other clinical trials during the course of this study.

Exclusion Criteria:

1. Known hypersensitivity or contraindication to progestins.
2. Abnormal Transvaginal Ultrasound (TVUS) or safety labs done during the screening period recognized as clinically significant by the investigator (or medically qualified designee).
3. Greater than 10% body weight change over previous year or planned significant weight loss during the study related to bariatric surgery, dieting or other causes.
4. Known or suspected current alcohol dependence syndrome, chronic marijuana use or any illicit drug use that may affect metabolism of the study product or study compliance.
5. Undiagnosed abnormal genital bleeding.
6. Undiagnosed vaginal discharge, lesions or abnormalities. Subjects diagnosed at screening with Chlamydia, or gonococcus infection may be included in the trial following treatment completion. In accordance with PI/medical designee assessment and local standards of practice, women with a history of genital herpes can be included if outbreaks are infrequent. Antiviral prophylactic therapy is permitted.
7. Uncontrolled thyroid disorder.
8. Current use of hormonal contraception including hormonal intrauterine device.
9. Use of a long-acting injectable hormonal contraceptive (e.g., cyclofem or depomedroxyprogesterone acetate) within the past 9 months prior to enrollment unless the subject has had at least one spontaneous menstrual cycle (at least two menses) since the last injection.
10. Recent use of hormonal oral, patch, intravaginal or intrauterine contraception unless that subject has had at least one complete menstrual cycle (at least two menses) since discontinuation before the treatment injection.
11. Women who are breastfeeding or are within 30 days of discontinuing breastfeeding unless the subject has already had a menses following discontinuation of breastfeeding.
12. Women planning to undergo major surgery during study participation.
13. Women planning pregnancy during their anticipated months of study participation.
14. Women who smoke > 15 cigarettes per day or who use >1 ml/day of nicotine-containing liquid for electronic cigarette must be evaluated by the PI for inclusion based on risk factors that would increase their risk for cardiovascular disease (CVD) and thromboembolism.
15. Current or past deep vein thrombophlebitis or thromboembolic disorders.
16. Known history of thrombophilia.
17. Cerebrovascular or cardiovascular disease or increased risk for arterial thrombosis.
18. Known or suspected carcinoma of the breast, endometrium, or any other known or suspected progestin-dependent neoplasia.
19. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive, unless she is stable on antidepressant medication.
20. Have a current need for exogenous hormones or therapeutic anticoagulants.
21. History of any other carcinoma (excluding basal cell carcinomas) unless in remission for more than 5 years.
22. Active liver disease or screening LFTs greater than twice the upper limit or normal.
23. Diastolic blood pressure (DBP) > 95 and Systolic blood pressure (SBP) > 145 mm Hg.
24. Clinically significant abnormal serum chemistry or hematology values according to the Principal Investigator's judgment.
25. Participation in another clinical trial involving an investigational drug or device within last the three months before treatment injection or planning to participate in another clinical trial during this study.
26. A Z-Score of ≤ -2.0 on baseline Dual-energy X-ray absorptiometry (DXA) scan (within 90 days prior to the injection visit).
27. Known HIV infection.
28. Women who use any medications on the Exclusionary Medication List (see Appendix 2) OR have used any within 90 days prior to the Injection visit.
29. Have issues or concerns (in the judgement of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.
30. Have known hypersensitivity to the active substance LB or any of the excipients of the study treatment.
31. Use any medications that can interfere with the metabolism of hormonal contraceptives, antibiotics that can interfere with metabolism of hormonal contraceptives, or any drugs designated by the FDA as falling in the Pregnancy and Lactation narrative subsections (formerly Category D or X medications).
32. Have previously participated in the study. A waiver may be requested to allow subjects to re-enroll, but only in a separate stage from the prior enrollment(s). Subjects must have had clear documentation of ovulation based on a rise in progesterone in their previous enrollment.
33. Be a site staff member with delegated study responsibilities or a family member of, or have a close relationship with, a site staff member with delegated study responsibilities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 136 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Measurement of levonorgestrel serum concentrations | 0, 2, 4, 6, 8, 24, 48, 96, 168, and 240 hours. Then weekly for up to 26 weeks.

SECONDARY OUTCOMES:
Ultrasound measurements of ovarian follicular development and ovulation including follicle diameter, total number of follicles, and the number of follicles exceeding a pre-specified threshold | Weekly up to 26 weeks
Measurement of Endometrial thickness | Weekly up to 26 weeks
Steroid hormone (Estradiol) concentration | Weekly up to 26 weeks
Gonadotropin (Follicle Stimulating Hormone and Luteinizing Hormone) concentrations | Weekly up to 26 weeks
Sex Hormone Binding Globulin (SHGB) concentration | Weekly up to 26 weeks
Bleeding patterns (spotting and light, moderate or heavy bleeding) reported through weekly subject diaries | Weekly up to 26 weeks
Side effects of LB as measured by adverse events reported | Weekly up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (7):
- United States (7):
  - University of California, Davis, Davis, California
  - Comprehensive Women's Health Center, Denver, Colorado
  - Boston Medical Center Corporation, Boston, Massachusetts
  - Columbia University, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No